CLINICAL TRIAL: NCT06850428
Title: Examining the Relationship Between Physical Activity Levels and Chronotype Tendencies in Individuals With Alcohol Dependence
Status: Recruiting | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Özge Çoban, Assistant Professor, Saglik Bilimleri Universitesi
Other Study IDs: 2025-116
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Abuse/Dependence
Keywords: chronotype; Alcohol abuse/Dependence; physical activity; physical activity level
MeSH Terms: conditions — Alcoholism; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Evening Type: This group includes individuals who are most productive in the evening. They prefer to stay awake until late in the evening and have difficulty getting up in the morning. They reach their highest energy levels and efficiency in the evening hours.
- Intermediate Type: This group is located between morning and evening types and includes individuals who can be productive at any time of the day. They neither have difficulty waking up early in the morning nor staying awake until late hours. They have a balanced energy level throughout the day.
- Morning type: This group includes individuals who have their highest energy levels in the morning hours. They wake up early in the morning and are most productive mentally and physically in the early hours of the day. It is generally preferred to start activities in the morning and sleep early.

SUMMARY:
Alcohol use disorders are characterized by excessive alcohol consumption and loss of control and are associated with high mortality and disease burden. The relationship between physical activity and alcoholism is complex, and low physical activity has been shown to be linked to alcohol consumption. Additionally, individuals' circadian rhythms (chronotypes) may influence alcohol consumption habits; Evening-type individuals are more likely to consume alcohol. This study aims to examine the relationship between physical activity levels and chronotype trends in individuals with alcohol addiction.

DETAILED DESCRIPTION:
This study aims to examine the relationship between physical activity levels and chronotype tendencies in individuals with alcohol dependency. Alcohol use disorders are characterized by excessive alcohol consumption and loss of control, and are associated with high mortality rates and disease burden. The relationship between physical activity and alcoholism is complex, with connections found between low physical activity levels and increased alcohol consumption. Additionally, individuals' circadian rhythms (chronotypes) can influence alcohol consumption habits, and evening-type individuals may be more likely to consume alcohol.

Participants and Method The study will include individuals aged 18-65, diagnosed with alcohol dependency according to DSM-5 criteria, and who have been in remission for at least one month. Individuals with active psychiatric disorders or physical disabilities will be excluded from the study. The sample size was determined using G*Power analysis, with a target of 207 participants for the ANOVA test. Participants will be reached through social media, support groups, rehabilitation centers, and health professionals, and assessments will be conducted via Google Forms. Participants will provide informed consent prior to participation. The sampling method is non-probability sampling.

Assessment Tools Chronotype Evaluation: The participants' circadian rhythms will be assessed using the "Morningness-Eveningness Questionnaire" in Turkish, which has proven validity and reliability. This scale consists of 19 items used to determine whether individuals have a morning, evening, or intermediate chronotype. Total scores will be categorized into five different chronotype groups based on predetermined ranges.

Physical Activity Level Evaluation The "International Physical Activity Questionnaire - Short Form," with proven validity in Turkish, will be used. This questionnaire measures walking, moderate, and vigorous physical activities and determines the total physical activity level in MET-minutes.

This research aims to contribute to a better understanding of the relationship between physical activity and chronotype in individuals with alcohol dependency. This study is designed as a cross-sectional observational research.

ELIGIBILITY:
Inclusion Criteria:

* Age: Being between 18-65 years old.
* Alcohol Dependence: Having alcohol dependence and this condition being confirmed according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria or stated based on self-report.
* Remission Status: Being in remission for at least 1 month (i.e., no active alcohol use).

Exclusion Criteria:

* Active Psychiatric Diseases: For example, individuals with active psychiatric diseases such as schizophrenia or bipolar disorder will not be included in the study.
* Physical Disability: Individuals with any physical disability will also be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 207
Sampling Method: Non-Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Relationship between physical activity levels and chronotype trends | from April 2025 to June 2025
  The main goal of the study is to determine the relationship between the participants' chronotypes (close to morning, intermediate type, close to evening type) and their physical activity levels in individuals with alcohol addiction.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Gülhane Faculty of Physiotherapy and Rehabilitation, Ankara, Keçiören, Turkey (Türkiye)